CLINICAL TRIAL: NCT01510158
Title: A Phase 3 Randomized, Double-Blind, Multicenter, Placebo-Controlled, Combination Study to Evaluate the Efficacy and Safety of Lesinurad and Allopurinol Compared to Allopurinol Alone in Subjects With Gout Who Have Had an Inadequate Hypouricemic Response to Standard of Care Allopurinol.
Brief Title: Combining Lesinurad With Allopurinol in Inadequate Responders
Acronym: CLEAR 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDEA594-301
Record Dates: First submitted 2012-01-11; First posted 2012-01-13 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lesinurad 200 mg + allopurinol (Experimental)
  Interventions: Drug: Lesinurad; Drug: Allopurinol
- lesinurad 400 mg + allopurinol (Experimental)
  Interventions: Drug: Lesinurad; Drug: Allopurinol
- Placebo + allopurinol (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Allopurinol

INTERVENTIONS:
Drug: Lesinurad — Tablets, 200 mg once daily (qd)
  Arms: lesinurad 200 mg + allopurinol
Drug: Lesinurad — Tablets, 400 mg qd
  Arms: lesinurad 400 mg + allopurinol
Drug: Placebo — Tablets, Placebo qd
  Arms: Placebo + allopurinol
Drug: Allopurinol — Tablets, ≥ 300 mg QD (≥ 200 mg qd for subjects with moderate renal impairment)
  Arms: lesinurad 200 mg + allopurinol
Drug: Allopurinol — Tablets, ≥ 300 mg QD (≥ 200 mg qd for subjects with moderate renal impairment)
  Arms: lesinurad 400 mg + allopurinol
Drug: Allopurinol — Tablets, ≥ 300 mg QD (≥ 200 mg qd for subjects with moderate renal impairment)
  Arms: Placebo + allopurinol

SUMMARY:
This study that compare the serum uric acid lowering effects, clinical benefits, and safety of lesinurad in combination with allopurinol to allopurinol alone in subjects with gout who have had an inadequate response to allopurinol.

DETAILED DESCRIPTION:
Allopurinol is the standard of care for the treatment of gout. Nevertheless, most patients treated with allopurinol do not achieve the recommended serum urate (sUA) target of < 6.0 mg/dL and need additional therapy to achieve the target. Probenecid and benzbromarone are uric acid transporter 1 (URAT1) inhibitors, generally recommended as second-line agents for patients who are either resistant to or intolerant of allopurinol. However, benzbromarone is not available in the US and probenecid is rarely used. Consequently, there is a clear unmet medical need for a new safe and effective therapy for gout, such as lesinurad, a potent URAT1 inhibitor, that can be used in combination with allopurinol in patients not responding adequately to allopurinol monotherapy so that very high rates of response can be achieved by nearly all gout patients, rather than a minority.The subjects selected for this study will have moderate to severe gout with an inadequate response to allopurinol

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures, the risks involved and willing to provide written informed consent before the first study related activity.
* Subject meets the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has been taking allopurinol as the sole urate-lowering therapy indicated for the treatment of gout for at least 8 weeks prior to the Screening Visit at a stable, medically appropriate dose, as determined by the investigator, of at least 300 mg per day (at least 200 mg for subjects with moderate renal impairment).
* Subject must be able to take gout flare prophylaxis with colchicine or an Nonsteroidal anti-inflammatory drug (NSAID) (including Cox-2 selective NSAID) ± PPI.
* Subject has an sUA level ≥ 6.5 mg/dL at the Screening Visit and ≥ 6.0 mg/dL at Day -7 Visit.
* Subject has reported at least 2 gout flares in the prior 12 months.
* Body mass index (BMI) < 45 kg/m2

Exclusion Criteria:

* Subject with known hypersensitivity or allergy to allopurinol.
* Subject who is taking any other approved urate-lowering medication that is indicated for the treatment of gout other than allopurinol within 8 weeks of the Screening Visit.
* Subject who is pregnant or breastfeeding.
* Subject who consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
* Subject with a history or suspicion of drug abuse within the past 5 years.
* Subject that requires or may require systemic immunosuppressive or immunomodulatory treatment.
* Subject with known or suspected human immunodeficiency virus (HIV) infection.
* Subject with a positive test for active hepatitis B or hepatitis C infection.
* Subject with a history of malignancy within the previous 5 years with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia or treated in situ Grade 1 cervical cancer.
* Subject within the last 12 months with: unstable angina, New York Heart Association class III or IV heart failure, myocardial infarction, stroke, or deep venous thrombosis; or subjects currently receiving anticoagulants.
* Subject with uncontrolled hypertension.
* Subject with an estimated creatinine clearance < 30 mL/min.
* Subject with active peptic ulcer disease requiring treatment.
* Subject with a history of xanthinuria, active liver disease, or hepatic dysfunction.
* Subject receiving chronic treatment with more than 325 mg of salicylates per day.
* Subject taking valpromide, progabide, or valproic acid.
* Subject who has received an investigational therapy within 8 weeks or 5 half-lives (whichever is longer) prior to the Screening Visit.
* Subject with any other medical or psychological condition, which might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Ardea Biosciences, Inc.
Locations (142):
- United States (142):
  - Athens, Alabama
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Mobile, Alabama
  - Pinson, Alabama
  - Glendale, Arizona
  - Goodyear, Arizona
  - Little Rock, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Tuscon, Arizona
  - Little Rock, Arkansas
  - Covina, California
  - Glendale, California
  - Huntington Beach, California
  - Inglewood, California
  - Lancaster, California
  - Lincoln, California
  - Orange, California
  - Sacramento, California
  - San Leandro, California
  - Santa Maria, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Milford, Connecticut
  - New London, Connecticut
  - Brooksville, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - East Bradenton, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Conyers, Georgia
  - Johns Creek, Georgia
  - Marietta, Georgia
  - Newnan, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Evansville, Indiana
  - Franklin, Indiana
  - La Porte, Indiana
  - Cedar Rapids, Iowa
  - Shawnee, Kansas
  - Elizabethtown, Kentucky
  - Paducah, Kentucky
  - Eunice, Louisiana
  - Metairie, Louisiana
  - Monroe, Louisiana
  - Natchitoches, Louisiana
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Southfield, Michigan
  - Traverse City, Michigan
  - Jackson, Mississippi
  - Florissant, Missouri
  - Hazelwood, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Missoula, Montana
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Endwell, New York
  - New York, New York
  - Syracuse, New York
  - Williamsville, New York
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Shelby, North Carolina
  - Tabor City, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Dayton, Ohio
  - Perrysburg, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Ashland, Oregon
  - Altoona, Pennsylvania
  - Belle Vernon, Pennsylvania
  - Clairton, Pennsylvania
  - Duncansville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Wexford, Pennsylvania
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Myrtle Beach, South Carolina
  - Rock Hill, South Carolina
  - Spartanburg, South Carolina
  - Brentwood, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Kingwood, Texas
  - Nassau Bay, Texas
  - Plabo, Texas
  - Plano, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Sealy, Texas
  - Waco, Texas
  - Bountiful, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Chesapeake, Virginia
  - Manassas, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Virginia Beach, Virginia
  - Port Orchard, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin

REFERENCES:
- [Derived] Topless R, Noorbaloochi S, Merriman TR, Singh JA. Change in serum urate level with urate-lowering therapy initiation associates in the immediate term with patient-reported outcomes in people with gout. Semin Arthritis Rheum. 2022 Oct;56:152057. doi: 10.1016/j.semarthrit.2022.152057. Epub 2022 Jun 29. PMID 35835008
- [Derived] Saag KG, Fitz-Patrick D, Kopicko J, Fung M, Bhakta N, Adler S, Storgard C, Baumgartner S, Becker MA. Lesinurad Combined With Allopurinol: A Randomized, Double-Blind, Placebo-Controlled Study in Gout Patients With an Inadequate Response to Standard-of-Care Allopurinol (a US-Based Study). Arthritis Rheumatol. 2017 Jan;69(1):203-212. doi: 10.1002/art.39840. PMID 27564409
- See also: Related Info — http://www.gouttrial.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lesinurad 200 mg + Allopurinol: lesinurad 200 mg qd plus allopurinol
- Lesinurad 400 mg + Allopurinol: lesinurad 400 mg qd plus allopurinol
- Placebo + Allopurinol: placebo qd plus allopurinol
Period: Overall Study
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Started | 202 | 203 | 202
Completed | 151 | 150 | 152
Not Completed | 51 | 53 | 50
Not completed — Adverse Event | 7 | 8 | 5
Not completed — Gout flare | 1 | 0 | 0
Not completed — Protocol Violation | 17 | 16 | 24
Not completed — Sponsor terminated study. | 2 | 0 | 2
Not completed — Lost to Follow-up | 13 | 16 | 9
Not completed — Withdrawal by Subject | 10 | 13 | 10
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol | Total
Number analyzed (Participants) | 201 | 201 | 201 | 603
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (10.7) | 52.3 (11.5) | 51.7 (11.7) | 51.9 (11.3)
Age, Customized [Number; unit: Participants]
  <65 | 181 | 168 | 169 | 518
  >=65 | 20 | 33 | 32 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 12 | 36
  Male | 192 | 186 | 189 | 567
Region of Enrollment [Number; unit: Participants]
  United States | 201 | 201 | 201 | 603

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With an sUA Level That is < 6.0 mg/dL
Time Frame: 6 Months, analysis after all subjects complete 12 months
Population: Intent-to-Treat Population
Measure: Number; unit: Proportion of Subjects
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Number analyzed (Participants) | 201 | 201 | 201
Proportion of Subjects | 0.542 | 0.592 | 0.279
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.26, 95% CI 2-sided [0.17 to 0.36], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.31, 95% CI 2-sided [0.22 to 0.41], Standard Error of Mean 0.05

2. Secondary Outcome: Gout Flares
Description: Mean rate of gout flares requiring treatment for the 6-month period from the end of Month 6 to the end of Month 12
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Gout Flares
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Number analyzed (Participants) | 201 | 201 | 201
Gout Flares | .60 (1.2) | .50 (1.2) | .60 (1.3)
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.9796, Negative Binomial Regression; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.61 to 1.61]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.6125, Negative Binomial Regression; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.54 to 1.43]

3. Secondary Outcome: Tophus
Description: Proportion of subjects with ≥ 1 target tophus at Baseline who experience complete resolution of at least 1 target tophus by Month 12
Time Frame: 12 Months
Measure: Number; unit: Proportion of Subjects
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Number analyzed (Participants) | 18 | 19 | 17
Proportion of Subjects | 0 | 0.211 | 0.294
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.0183, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.29, 95% CI 2-sided [-0.51 to -0.08]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.5974, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.08, 95% CI 2-sided [-0.37 to 0.2]

ADVERSE EVENTS:
Description: Overall number of baseline participants used to determine number of participants at risk.
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Serious Adverse Events (participants affected / at risk) | 9/201 | 16/201 | 11/201
Other Adverse Events (participants affected / at risk) | 147/201 | 156/201 | 138/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Allopurinol (N=201) | Lesinurad 400 mg + Allopurinol (N=201) | Placebo + Allopurinol (N=201)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (2)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Allopurinol (N=201) | Lesinurad 400 mg + Allopurinol (N=201) | Placebo + Allopurinol (N=201)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness transitory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Androgen deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular icterus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (3) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 8 (8) | 8 (8)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 9 (11) | 9 (9)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 6 (6) | 5 (5)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 3 (3) | 5 (5)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 5 (5) | 3 (4)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 5 (7) | 2 (2) | 3 (3)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 6 (6) | 5 (6)
Pain (General disorders) | 3 (3) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 5 (6) | 6 (6) | 6 (6)
Secretion discharge (General disorders) | 1 (2) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2) | 4 (4)
Abscess limb (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 7 (8) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 5 (5) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 4 (5) | 3 (3) | 4 (4)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (6) | 6 (6) | 8 (10)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 17 (23) | 15 (18) | 14 (17)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (3) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peptostreptococcus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 9 (11) | 12 (15) | 4 (4)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 22 (28) | 18 (22) | 11 (13)
Urinary tract infection (Infections and infestations) | 3 (3) | 10 (10) | 4 (5)
Viral infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 7 (10) | 6 (6)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 6 (7) | 8 (9)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 2 (2)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 10 (10) | 10 (12) | 7 (9)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood amylase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood bicarbonate decreased (Investigations) | 3 (4) | 5 (7) | 3 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 9 (10) | 16 (16) | 5 (5)
Blood creatinine increased (Investigations) | 7 (11) | 14 (19) | 2 (2)
Blood glucose increased (Investigations) | 4 (5) | 4 (4) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood testosterone decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 6 (6) | 4 (4)
Blood urea increased (Investigations) | 2 (4) | 3 (4) | 2 (2)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (1)
Body temperature decreased (Investigations) | 1 (4) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (6)
Glucose urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haematocrit increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitamin b12 decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 0 (0)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 16 (18) | 19 (23)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 9 (12) | 19 (21)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 9 (10)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8) | 4 (4)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5) | 9 (11)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cataplexy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 9 (9) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (9) | 12 (15) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (5)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 2 (2) | 4 (4)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 4 (4) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 4 (4) | 4 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Urethral perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 4 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (5) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 7 (7) | 7 (7)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.